CLINICAL TRIAL: NCT03886246
Title: Effisayil™ ON: An Open-label, Long Term Extension Study to Assess the Safety and Efficacy of Spesolimab Treatment in Patients With Generalized Pustular Psoriasis (GPP)
Brief Title: Effisayil™ ON: A Study to Test Long-term Treatment With Spesolimab in People With Generalized Pustular Psoriasis Who Took Part in a Previous Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0025; 2018-003080-56 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Spesolimab (every 6 weeks) (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab (every 12 weeks) (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab (every 4 weeks) (Experimental)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Solution for infusion
  Arms: Spesolimab (every 6 weeks)
Drug: Spesolimab — Solution for injection

SUMMARY:
This study is open to people with generalized pustular psoriasis (GPP). People can only take part if they have completed treatment in a previous study with spesolimab (1368-0013 or 1368-0027).

The goal of this study is to find out how well people with GPP tolerate long-term treatment with spesolimab. The study also tests whether spesolimab helps improve GPP symptoms and how quickly the symptoms improve after a flare-up.

Every participant gets spesolimab for almost 5 years (252 weeks). Depending on their symptoms and whether they had a GPP flare during the previous trial, they get spesolimab every few weeks. When participants have a GPP flare during this trial, they get spesolimab as an infusion into a vein.

Participants visit their doctors regularly. During these visits, the doctors collect information on any health problems of the participants. To assess the study endpoints, doctors regularly check participants' skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who have completed the treatment period without premature discontinuation in the previous spesolimab trial and are willing and able to continue treatment in the current trial
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in Section 4.2.2.3 as well as in the patient information. Note: A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is not a method of permanent sterilization. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Signed and dated written informed consent and assent for the current trial 1368-0025, in accordance with ICH-GCP and local legislation prior to admission to the current trial

Exclusion Criteria:

* Evidence of flare symptoms of moderate/severe intensity at screening.
* Treatment with any restricted medication as specified in the protocol, or any drugs considered by the investigator likely to interfere with the safe conduct of the study since the last visit of the previous spesolimab trial and during the screening period for the current trial, with the exception of methotrexate, cyclosporine, or retinoids started following rescue treatment for GPP flare in trial 1368-0027.
* Severe, progressive, or uncontrolled hepatic disease, defined as >3- fold Upper Limit of Normal (ULN) elevation in Aspartate Transaminase (AST) or Alanine Aminotransferase (ALT) or alkaline phosphatase, or >2- fold ULN elevation in total bilirubin.
* Patients with congestive heart disease, as assessed by the investigator.
* Relevant chronic or acute infections including human immunodeficiency virus (HIV) or viral hepatitis. A patient can be re-screened if the patient was treated and is cured from acute infection.
* Active or Latent tuberculosis (TB):

  * Patients with active tuberculosis should be excluded
  * Patients will be screened with Interferon Gamma Release Assay (IGRA) such as QuantiFERON®-TB-Gold Plus or T-spot®. Patients with positive IGRA (indicating active or latent tuberculosis) are excluded unless they have completed treatment for active or latent tuberculosis per investigator discretion, at the time of screening.
  * Patients with indeterminate QuantiFERON®-TB-Gold Plus or invalid/borderline T-spot® may be retested with IGRA (once) or Tuberculin Skin test (TST).
  * TST or any alternative test/procedure (as per local standards) to rule out TB can be performed if IGRA is not available or indeterminate. A TST reaction ≥10mm (≥5mm if receiving ≥15mg/d prednisone or other immunosuppressant) is considered positive. Patients with a positive TST are excluded unless they have completed treatment as above.
* History of allergy/hypersensitivity to a systemically administered trial medication agent or its excipients.
* Any documented active or suspected malignancy at screening, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix.

Further exclusion criteria apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-04-27 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs) up to week 252 of maintenance treatment | Up to 252 Weeks

SECONDARY OUTCOMES:
The reoccurrence of a GPP flare defined by GPPGA | Up to 252 Weeks
  The total GPPGA score ranges from 0 to 4 with a higher score indicating a higher grade of inflammation.
Time to first achievement of a GPPGA score of 0 or 1 (Patients received flare rescue Treatment) | Up to 252 Weeks
A GPPGA pustulation sub-score of 0 indicating no visible pustules, by visit | Up to 252 Weeks
Change from baseline in Psoriasis Symptom Scale (PSS) score, by visit | Up to 252 Weeks
  The PSS score ranges from None to Very Severe with a higher score indicating a higher severity of psoriasis symptom.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (2):
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
- Hospital Italiano de Buenos Aires, CABA, Argentina
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Clínica Dermacross S.A., Vitacura, Chile
- China (5):
  - Sun yet-sen Memorial Hospital, Sun yet-sen Univesity, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Shanghai Skin Disease Hospital, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
- France (4):
  - HOP Saint-André, Bordeaux
  - HOP l'Archet, Nice
  - HOP Saint-Louis, Paris
  - HOP Robert Debré, Reims
- Germany (7):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite Universitätsmedizin Berlin KöR, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum der Universität München - Campus Innenstadt, München
  - Westfälische Wilhelms-Universität Münster, Münster
  - Klinikum Oldenburg AöR, Oldenburg
- Istituto Clinico Humanitas, Rozzano (MI), Italy
- Japan (4):
  - Nagoya City University Hospital, Aichi, Nagoya
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki, Inashiki-gun
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
- Malaysia (9):
  - Hospital Pulau Pinang-Pulau Pinang-21953, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Sultan Ismail, Johor Bahru
  - Queen Elizabeth Hospital-Kota Kinabalu-40735, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Pakar Sultanah Fatimah, Muar town
- Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Mexico
- Philippines (3):
  - Southern Philippines Medical Center -Davao-62091, Davao City
  - Iloilo Doctors Hospital, Iloilo City, Iloilo
  - Center for Skin Research, Testing and Product Development, Makati City
- Russia (5):
  - SBHI Chelyabinsk Reg.Clin.Derma.Dispen., Chelyabinsk
  - LLC "Medical Center Azbuka Zdorovia", Kazan'
  - FSBEI HE "Kirov State Medical University", Kirov
  - LLC Skin Disease Clinic of Pier Volkenstein, St. Petersburg, Saint Petersburg
  - Saratov State Med.Univ.n.a.Razumovskogo, Saratov
- Singapore General Hospital, Singapore, Singapore
- Severance Hospital, Seoul, South Korea
- Hospital Sant Joan de Déu, Esplugues Del Llobregat, Spain
- Taiwan (2):
  - Chang Gung Medical Foundation (CGMF) - Linkou Bran, Linkou District
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Institute of Dermatology, Bangkok
  - Ramathibodi Hospital, Bangkok
- Tunisia (3):
  - Farhat Hached Hospital, Sousse
  - La Rabta Hospital, Tunis
  - Hedi Chaker Hospital, Department of Dermatology, Tunisia
- Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul, Turkey (Türkiye)
- Vietnam (2):
  - National Hospital of Dermatology and Venereology, Hà Nội
  - HCMC Hospital of Dermato-Venereology-Ho Chi Minh-66092, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/